CLINICAL TRIAL: NCT03528980
Title: Comparing the Impact of Weight Loss Induced by Bariatric Surgery or Through a Standard Nutritional Management on Sexual Function and Sperm Quality in Men With Severe Obesity - Multicenter, Prospective
Brief Title: Impact of Weight Loss Induced by Bariatric Surgery or Nutritional Management on Sexual Function in Men With Severe Obesity
Acronym: SexOb
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2011_07; 2011-A01012-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-04-25; First posted 2018-05-18 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2021-03

CONDITIONS: Obesity; Bariatric Surgery Candidate
Keywords: fertility; bariatric surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bariatric surgery
- standard nutritional management

SUMMARY:
Study of the impact of weight loss induced by surgery (interventional group) or optimal nutritional management (control group) on sexual function in men with severe obesity

ELIGIBILITY:
Inclusion Criteria:

* Severe obesity with BMI> 25 kg / m2

Exclusion Criteria:

* Patient having undergone sterilization

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: patients with morbid obesity,
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Improvement of sexual function assessed by International Index for Erectile Dysfunction (IIED) | at 1 year
  This questionnaire consists of 15 questions addressing the following topics: erectile function, orgasmic function, sexual desire, satisfaction of the sexual relation, satisfaction of the relationship in general. Each question is scored from 0 to 5. All responses are scored between 0 and 75. Sexual function is considered normal if the IIED score is greater than 25

SECONDARY OUTCOMES:
Percentage of patients with normal sexual function (IIED> 25) with and without surgery. | ay 1 year
Change the spermatic parameters before and after weight loss in both groups | at 1 year and 2 years
Change the serum profile of sex hormones before and after weight loss in both groups a | at 1 year
Correlate the spermatic profile to the different nutritional deficiencies high lighted after the bariatric surgery | at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Caiazzo, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (3):
- France (3):
  - Chu de Caen Normandie, Caen
  - CHRU, Hôpital Claude Huriez, Lille
  - Chu Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No